CLINICAL TRIAL: NCT04781803
Title: Cyclosporine on Day Zero as Prophylaxis for Cytokine Release Syndrome in Outpatient Haploidentical Hematopoietic Stem Cell Transplantation
Brief Title: Cyclosporine on Day Zero as Prophylaxis for Cytokine Release Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, David Gomez Almaguer, Chief of service, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HE21-00003
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Stem Cell Transplant Complications; Cytokine Release Syndrome
Keywords: Cyclosporin; Haploidentical; Outpatient
MeSH Terms: conditions — Cytokine Release Syndrome | interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Cyclosporine 6 mg/kg orally divided into two doses per day starting in the morning on day 0 after transplantation, mycophenolic acid 1 gram orally (2 tablets 500 mg) from day 0 post-transplant and PT-CY at 50 mg/kg per day on day +3 and +4.
  Interventions: Drug: Cyclosporine
- Arm 2 (No Intervention): Cyclosporine 6 mg/kg orally divided into two doses per day starting in the morning on day +5 of the transplant, mycophenolic acid 1 gram orally (2 tablets of 500 mg) from day +5 post-transplant and post-transplant cyclophosphamide (PT-CY) at 50 mg/kg per day on days +3 and +4

INTERVENTIONS:
Drug: Cyclosporine — Cyclosporine 6 mg/kg and mycophenolic acid 1 gram orally on day 0 post-transplant
  Arms: Arm 1

SUMMARY:
Phase II, randomized controlled, unblinded clinical trial. Will evaluate whether the administration of oral cyclosporine started on day 0 of transplantation is effective in reducing the incidence of cytokine release syndrome (CRS) in patients who receive an outpatient haploidentical transplant.

DETAILED DESCRIPTION:
CRS is usually limited after the administration of post-transplant cyclosporine (PT-CsA) administered on days +3 and +4, however, there is no standard prevention or treatment regimen for CRS after haplo-TCPH and therapeutic behavior has usually been adopted.

Sample of 32 patients between the ages of 16 and 60 who receive their first haploidentical transplant at our center. In the control group, CsA 6 mg/kg orally divided into two doses per day starting in the morning on day +5 of the transplant, mycophenolic acid 1 gram orally (2 tablets of 500 mg) from day +5 post-transplant and post-transplant cyclophosphamide (PT-CY) at 50 mg/kg per day on days +3 and +4 and in the experimental group, CsA 6 mg/kg orally divided into two doses per day starting in the morning on day 0 after transplantation, mycophenolic acid 1 gram orally (2 tablets 500 mg) from day 0 post-transplant and PT-CY at 50 mg/kg per day on day +3 and +4.

Will document the presence of CRS and its degree, as well as the need for hospitalization, associated infectious processes, and a day to recover neutrophils and platelets. Additionally, 4 blood samples will be taken from the patients to determine the level of cytokines and C-reactive protein.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 16-60 years of age who receive their first haploidentical transplant.

Exclusion Criteria:

* Patients positive for the human immunodeficiency virus (HIV), Hepatitis B or C virus
* Pregnancy or lactation
* Patients with documented infection at the time of transplantation
* Presence of previous autoimmune diseases
* Inability to tolerate the oral route

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-03-25 (Estimated); Primary Completion 2023-01-17 (Estimated); Study Completion 2023-02-17 (Estimated)

PRIMARY OUTCOMES:
Cytokine Release Syndrome | day 0 to day 30
  Presence of Fever, hypotension, hypoxemia

CONTACTS AND LOCATIONS:
Overall Officials: Oscar González-Llano, MD, Principal Investigator — Hospital Universitario ¨Dr. José Eleuterio González
Locations (1):
- Hospital Universitario Dr. José E. González, Centro Universitario contra el Cáncer, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No